CLINICAL TRIAL: NCT06121557
Title: Phase I Study of Autologous Tumor-Draining Lymph Node-Derived Lymphocytes for Advanced HER2-Negative Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Erwei Song, M.D., Ph.D., Director of Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2021] 03-01
Record Dates: First submitted 2023-10-26; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Breast Neoplasms
Keywords: HER2-Negative; Lymph Node; Lymphocytes; Adoptive Cell Therapy; Camrelizumab; Chemotherapy; Antibody-Drug Conjugate; Poly(ADP-ribose) Polymerase Inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — Surgical Procedures, Operative; Cyclophosphamide; fludarabine; Interleukin-2; camrelizumab; arginine decarboxylase; Poly(ADP-ribose) Polymerase Inhibitors

STUDY DESIGN:
Intervention Model Description: Single-arm, dose-escalation and dose-expansion study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LNL treatment + Camrelizumab + another anti-tumor drug (Experimental): Participants receive LNL treatment, which consists of non-myeloablative lymphocyte depleting regimen of chemotherapy with cyclophosphamide and fludarabine, followed by infusion of LNL and interleukin-2. After LNL treatment, participants receive camrelizumab PLUS another anti-tumor drug chosen from chemotherapeutic drug, ADC, or PARP inhibitor at investigator's discretion.
  Interventions: Procedure: Surgery for harvesting tumor-draining lymph nodes; Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Tumor-draining lymph node-derived lymphocyte (LNL); Biological: Interleukin-2; Biological: Camrelizumab; Drug: Chemotherapeutic drug, ADC or PARP inhibitor

INTERVENTIONS:
Procedure: Surgery for harvesting tumor-draining lymph nodes — A sample of the participant's tumor-draining lymph nodes will be collected and sent to the biotherapy center for LNL isolation and expansion.
Drug: Cyclophosphamide — Cyclophosphamide will be administered at 500 mg/m^2 IV daily for three days. Cyclophosphamide will be initiated five days prior to the anticipated LNL transfer, and the precise timing will depend on the rate of in vitro LNL growth.
Drug: Fludarabine — Fludarabine will be administered at 30 mg/m^2 IV daily for three days. Fludarabine will be initiated five days prior to the anticipated LNL transfer, and the precise timing will depend on the rate of in vitro LNL growth.
Biological: Tumor-draining lymph node-derived lymphocyte (LNL) — In the dose-escalation portion, participants receive ascending dose (1×10^9~18×10^9), single Infusion of LNL on day 0. In the dose-expansion portion, participants receive single infusion of LNL at the recommended phase 2 dose (RP2D).
  Other Names: LNL
Biological: Interleukin-2 — Eight to twelve hours after completing the LNL infusion, all participants will receive intermediate-dose decrescendo IL-2 IV.
  Other Names: IL-2
Biological: Camrelizumab — Camrelizumab will be administered at a dose of 200mg (3mg/kg for participants whose weight is below 50kg) IV on Day 1 of each 21-day cycle until unacceptable toxic effects or disease progression or other termination criteria appeared.
  Other Names: SHR-1210
Drug: Chemotherapeutic drug, ADC or PARP inhibitor — Another anti-tumor drug chosen from chemotherapeutic drug, ADC, or PARP inhibitor will be administered at investigator's discretion.

SUMMARY:
RATIONALE: Patients with HER2-negative advanced breast cancer have limited choice on targeted therapies, and often show only modest responses to available immunotherapies. Adoptive cell therapy with tumor-infiltrating lymphocytes has difficulties in preparing enough cells from solid tumors and overcoming the exhaustion and dysfunction of T cells, which limit its clinical use. Tumor-draining lymph node-derived lymphocytes (LNLs) that have abundant tumor-specific T cells, rather than exhausted T cells, are easier to produce. It is not yet known whether LNL treatment is safe and effective in patients with advanced HER2-negative breast cancer.

PURPOSE: This phase I trial is mainly to study the safety of autologous LNL in patients with advanced HER2-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for participation in this trial, the participant must:

1. Have signed the informed consent to study participation.
2. Be a female subject and aged between 18 and 70 years.
3. Have locally advanced or recurrent inoperable HER2-negative breast cancer (Stage IIIB~IIIC) which cannot be treated with curative intent OR have metastatic breast cancer (Stage IV). HER2-negative breast cancer is defined by the most recent ASCO/CAP guidelines. Participants should appear clinically stable in the opinion of the investigator.
4. Participants with estrogen receptor (ER)-positive and/or progesterone receptor (PR)-positive breast cancer have failed at least one line of hormonal therapy or CDK4/6 inhibitor, or are appropriate candidates for chemotherapy. Participants with ER-positive and/or PR-positive breast cancer may have received unlimited prior chemotherapy. Participants with triple-negative breast cancer (TNBC) may have received unlimited prior treatments for breast cancer.
5. Have not received any prior adoptive cell therapy.
6. Be suitable for treatment with camrelizumab and another anti-tumor drug chosen from chemotherapeutic drug, ADC, or PARP inhibitor as judged by the investigator.
7. Have accessible tumor-draining lymph nodes by surgery to grow LNL.
8. Have measurable disease based on RECIST 1.1. Target lesions situated in a previously irradiated area are considered measurable, only if they have shown unequivocal progression based on RECIST 1.1 after radiation therapy.
9. Have provided recently or newly obtained biopsy from a locally advanced or recurrent inoperable or metastatic tumor lesion for pathological examination of molecular subtype and PD-L1 expression, unless contraindicated due to site inaccessibility and/or participant safety concerns.
10. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
11. Have life expectancy ≥4 months.
12. Demonstrate adequate normal organ function:

    NOTE: Blood component or cytokine therapy is not allowed within 14 days before surgery.
    1. Routine blood test:

       * Absolute neutrophil count (ANC) ≥1.5×10^9/L
       * Lymphocyte count (LC) >0.5×10^9/L
       * Platelets (PLT) ≥100×10^9/L
       * Hemoglobin (Hb) ≥90 g/L
    2. Liver function test:

       * AST and ALT ≤2.5×ULN (≤5×ULN for participants with liver metastases)
       * ALP ≤2.5×ULN (≤5×ULN for participants with liver or bone metastases)
       * Total bilirubin ≤1.5×ULN (≤3.0 mg/dL for participants with Gilbert's syndrome)
    3. Renal function test:

       · Calculated creatinine clearance (CrCL) ≥45 mL/min OR creatinine ≤1.5×ULN
    4. Coagulation function test:

       * APTT ≤1.5×ULN
       * INR or PT ≤1.5×ULN
    5. Doppler echocardiography:

       · Left ventricular ejection fraction (LVEF) ≥50%
    6. Pulmonary function test:

       * FEV1 ≥60%
13. Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through one year (or longer as specified by local institutional guidelines) after the last dose of study treatment. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days prior to LNL infusion.
14. Have a specified washout period from prior anti-tumor therapies to the enrollment:

    * Angiogenesis inhibitors: 4 weeks
    * Chemotherapy or targeted therapy: 3 weeks
    * Radiotherapy: 2 weeks
    * Hormonal therapy: one week

Have recovered from prior therapy-related adverse events to Grade≤1 per CTCAE version 5.0 criteria or met the criteria of normal organ function specified above, except for second-degree peripheral nerve injury, alopecia, leukoderma, hypothyroidism controlled by thyroid hormone replacement therapy, type 1 diabetes controlled by insulin therapy, and other irreversible toxic events that would not be exacerbated by LNL infusion as judged by the investigator (e.g., hearing loss).

Exclusion Criteria:

The participant must be excluded from participating in this trial if the participant:

1. Has rapidly progressing tumors, as judged by the investigator.
2. Has known active CNS metastases and/or carcinomatous meningitis except for previously treated and radiographically stable CNS metastases, or CNS metastases without medication requirement and corticosteroid dependence. To demonstrate radiographic stability of brain metastases, a minimum of 2 post-treatment brain imaging assessments are required: (1) The first brain imaging must be acquired after treatment of brain metastases has been completed; (2) The second brain imaging must be obtained during screening and 4 weeks after the previous post-treatment brain imaging.
3. Has spinal cord compression not relieved by surgery or radiotherapy. Participants with previously treated spinal cord compression may participate provided that the compression-related symptoms are relieved within more than one week prior to surgery for tumor-draining lymph nodes.
4. Has uncontrolled pleural effusion, pericardial effusion or ascites. Participants with indwelling catheter may participate.
5. Has uncontrolled cancer pain as judged by the investigator. Participants requiring pain medication must have a treatment plan before enrollment. Symptomatic lesions suitable for palliative radiotherapy should be treated before enrollment.
6. Has a known additional malignancy that is progressing or requires active treatment within the last 5 years. Exceptions include basal or squamous cell carcinoma of the skin, and thyroid cancer that has undergone potentially curative therapy or in situ cervical cancer.
7. Has a known history of cardiovascular disease, including but not limited to, (1) congestive heart failure (New York Heart Association [NYHA] functional classification Class > 2), (2) unstable angina pectoris, (3) myocardial infarction in the past 3 months, (4) supraventricular arrhythmia or ventricular arrhythmia that requires treatments.
8. Has interstitial pneumonia or active pneumonia that has clinical implication, or other respiratory diseases that seriously affect pulmonary function.
9. Has an active infection requiring systemic therapy or has an unexplained fever of >38.5℃ except fevers caused by cancer.
10. Has arterial and/or venous thrombotic events in the past 5 months, e.g., cerebrovascular accident, deep vein thrombosis or pulmonary embolism.
11. Is currently participating in a clinical study and receiving an investigational agent and/or using an investigational device, or has participated in a clinical study and received an investigational agent and/or used an investigational device within 4 weeks prior to enrollment.

    Note: Subjects who have entered the follow-up phase of a clinical study may participate as long as 4 weeks have elapsed since the last dose of the investigational agent and/or removal of the device.
12. Has a known psychiatric, alcohol abuse or substance abuse disorders.
13. Is pregnant or breastfeeding.
14. Has an active autoimmune disease, a history of autoimmune disease, or autoimmune disease that has required systemic treatment (e.g., with use of prednisone at a dose of >10 mg per day or other corticosteroids at an equivalent dose). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is allowed.
15. Has a history of congenital immunodeficiency or acquired immunodeficiency (e.g., positive serology test for HIV).
16. Has tuberculosis in the past one year, or has a history of active tuberculosis more than one year but did not receive regular treatments.
17. Has known active hepatitis B or hepatitis C. Participants that are hepatitis B surface antigen (HBsAg) or hepatitis B core antigen (HBcAg) positive may participate provided that the HBV DNA level is normal. Participants that are hepatitis C antibody positive may participate provided that the HCV DNA level is normal. Carriers of HBV or HCV must receive anti-virus therapy, and take regular DNA copy number tests during this trial.
18. Has received a live vaccine within 4 weeks prior to enrollment, or plans to receive a live vaccine during this trial.
19. Has a history of allogeneic bone marrow or organ transplant.
20. Has a history of hypersensitivity or allergy to the drugs in this study and any of their components including but not limited to, LNL, cyclophosphamide, fludarabine, interleukin-2, dimethyl sulphoxide (DMSO), human serum albumin (HSA), dextran-40, antibiotics (β-lactam antibiotics, gentamicin), camrelizumab, or another anti-tumor drug that the investigator intends to choose.
21. Has contraindication for use of IL-2, including but not limited to, refractory or intractable epilepsy, and active gastrointestinal bleeding.
22. Has a history of Grade≥2 neuropathy.
23. Is receiving any medication prohibited in combination with study treatment as described in the respective product labels, unless medication was stopped within 7 days prior to enrollment.
24. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with participation for the full duration of the study, or render study participation not compatible with the participant's best interest, in the opinion of the investigator.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicity (DLT) | From the LNL infusion up to 28 days post-infusion
  Adverse events are reported based upon Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 criteria. DLT will be defined as a non-hematologic Grade 3 or higher adverse event, occurring within the 28 days immediately after LNL infusion, that is probably or definitely related to LNL infusion, and lasts more than 28 days or does not resolve to Grade<3 despite treatment with dexamethasone at 10 mg per 12 hours IV for 7 days (or other corticosteroid at equivalent dose), and/or tocilizumab at 8mg/kg IV for three times.
Incidence of Grade≥3 Treatment-Emergent Adverse Event (TEAE) | From the LNL infusion up to 28 days post-infusion
  Adverse events are reported based upon CTCAE version 5.0 criteria. The incidence of Grade≥3 TEAE occurring within the 28 days immediately after LNL infusion will be summarized with descriptive statistics.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately two years
  Objective response rate is defined as the percentage of participants in the analysis population who have achieved complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). The percentage of participants who experienced a CR or PR is presented.
Disease Control Rate (DCR) | Up to approximately two years
  Disease control rate is defined as the percentage of participants who have achieved CR or PR or have demonstrated stable disease (SD) for at least 24 weeks, per RECIST 1.1.
Duration of Response (DOR) | Up to approximately two years
  For participants who demonstrate a confirmed CR or confirmed PR per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) per RECIST 1.1 or death due to any cause, whichever occurs first.
Progression-Free Survival (PFS) | Up to approximately two years
  Progression-free survival is defined as the time from enrollment to the first documented PD per RECIST 1.1 or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately five years
  Overall survival is defined as the time from enrollment to death due to any cause. Participants without documented death at the time of the analysis were censored at the date of the last follow-up.
Levels of multiple different cytokines in blood samples before and after LNL infusion. | Up to approximately two years
  Levels of multiple different cytokines in blood samples including Granzyme B, IFN-γ, GM-CSF, IL-2, IL-4, IL-6, etc. will be measured using cytokine chips, ELISA or flow cytometry at various time points before and after LNL infusion.
Distribution of T cell subsets in blood samples before and after LNL infusion. | Up to approximately two years
  Distribution of T cell subsets in blood samples will be measured using flow cytometry at various time points before and after LNL infusion.
Distribution of T-cell receptor (TCR) clonotype in blood samples before and after LNL infusion. | Up to approximately two years
  Distribution of T-cell receptor (TCR) clonotype in blood samples will be measured using TCR sequencing at various time points before and after LNL infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Erwei Song, M.D., Ph.D., Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China